CLINICAL TRIAL: NCT06522373
Title: Phase I Trial of MT-0169 in CD38+ Acute Leukemia With Relapsed/Refractory or Measurable Residual Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0177; NCI-2024-06176 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-04

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Escalation Adults: MT-0169 (Experimental)
  Interventions: Drug: MT-0169
- Escalation Pediatrics: MT-0169 (Experimental)
  Interventions: Drug: MT-0169
- Expansion Adults: MT-0169 (Experimental)
  Interventions: Drug: MT-0169
- Expansion Pediatrics: MT-0169 (Experimental)
  Interventions: Drug: MT-0169

INTERVENTIONS:
Drug: MT-0169 — Given by Vein (IV)

SUMMARY:
To learn if MT-0169 is safe to give to patients with AML or T-ALL. The effects of this drug will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

To study the safety and tolerability of MT-0169.

Secondary Objectives:

To study preliminary efficacy of MT-0169 in terms of morphologic and MRD response rates and survival outcomes.

Exploratory Objectives:

To determine the plasma concentration and pharmacokinetic (PK) parameters of MT-0169.

To estimate proportion of MRD+ patients who achieved 1 log fold reduction in MRD burden.

To explore, additional response and survival outcomes, potential biomarkers of response, resistance and impact on immune microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients need to be ≥ 12 years of age.
2. ECOG performance status of o to 2.
3. Patients need to have a confirmed diagnosis of T-ALL, or AML, MDS/AML, (10% to 19% blasts), or mixed or biphenotypic leukemia, per the International Consensus Classification or the WHO classification.40,41
4. Patients need to have either relapsed or refractory disease: T-ALL, AML, MDS/AML, MPAL, biphenotypic leukemia; or patients with AML or T-ALL in CR/CRi/CRh with measurable residual disease (MRD), and no available standard or approved treatment options. Patients with MPAL or biphenotypic leukemia will only be eligible during the dose escalation phase.
5. Patients will need to have positive CD38 expression on leukemia cell population for dose escalation cohort and CD38 expression ≥20% on leukemia cell population by flow cytometry or IHC for dose expansion cohorts as assessed by standard of care flow cytometry.
6. Relapsed or refractory disease defined by standard criteria as follows

   a. Relapsed: Bone marrow blasts ≥5%, reappearance of blasts in the blood, or development of extramedullary disease following achievement of CR/CRi/MLFS b. Refractory: Failure to achieve CR/CRi/MLFS following initial treatment, with evidence of persistent leukemia by blood and/or bone marrow evaluation c. Patients with AML must have received appropriate prior therapy in order for patient to be deemed relapsed or refractory, including any of the following i. At least 1 cycle of purine analogue containing intensive induction chemotherapy regimen, e.g., FLAG-Ida, CLIA or CLAG-M or similar regimens with or without venetoclax.42,43 ii. At least 1 cycle of intensive induction chemotherapy with venetoclax, e.g., 7 + 3 or CPX-351 with venetoclax iii. At least 2 cycles of intensive induction chemotherapy such as 7 + 3 or 5 + 2 or similar regimens without venetoclax iv. 2 cycles of venetoclax with HMA/LDAC +/- other agents v. 4 cycles of HMA-based regimen d. Patients with T-ALL should have received at least 1 cycle of a standard or appropriate frontline regimen per NCCN or ELN2023 guidelines for ALL.44,45 e. Patients with mixed or biphenotypic leukemia should have received one AML or ALL type regimen as mentioned above f. Pediatric patients need to have R/R disease after at least one line of standard pediatric frontline regimen.
7. For patients in first relapse, the dose escalation cohort will only enroll patients in early first relapse, i.e., first remission duration of ≤12 months.

   1. Patients relapsing with persistent or new TP53 mutation will be eligible irrespective of CR1 duration.
   2. Older/unfit patients who relapse on venetoclax based maintenance regimen will be eligible irrespective of CR1 duration.
8. Patients without overt relapse but positive measurable residual disease (MRD) with a response status of composite CR (cCR = CR/CRi/CRh, i.e., <5% blasts) will be eligible for the trial

   1. Patients with AML will be eligible if they have MRD ≥ 0.1% using multiparametric flow cytometry assay.
   2. Patients with T-ALL will be eligible if they have MRD ≥0.01% by multiparametric flow cytometry, or PCR/NGS (i.e., ≥ 100 residual clonal cells per million nucleated cells evaluated by T-cell repertoire sequencing by PCR and/or NGS [commercial Adaptive clonoSEQ assay]).7,11
   3. Patients in 2nd or higher cCR for AML or T-ALL will be eligible after at least one cycle of salvage therapy.
   4. Patients with MRD relapse after allo-SCT or during consolidation or maintenance therapy will be eligible.
   5. Patients with AML in first remission cCR will be eligible if they have adverse risk AML per ELN2022 and must have received at least,

   i. 1 cycle of intensive induction and 1 cycle of consolidation chemotherapy with intermediate or high-dose cytarabine based regimen,46 or ii. 4 cycles of venetoclax-based lower intensity regimen containing HMA or LDAC, due to know adverse prognosis of such patients,22,23,47,48 or iii. 4 cycles of frontline HMA-based regimen (i.e., CR1), or f. Patients with T-ALL in first remission (CR1) will be eligible if they have positive MRD after 2 cycles of frontline therapy per NCCN or ELN2023 guidelines for ALL.44,45
9. Patients relapsing after allo-SCT may be eligible if they have recovered from all transplant-related toxicities, with no more than grade 1 chronic GVHD.
10. Patients with actionable mutations with FDA-approved therapies, e.g., FLT3, IDH1/2 inhibitors may be enrolled after they have received at least one appropriate line of available FDA approved treatment option.
11. Adequate hepatic function (direct bilirubin ≤ 2 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement, and AST and/or ALT ≤ 2.5 x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT ≤ 3 x ULN will be considered eligible.)
12. Adequate renal function with creatinine clearance ≥ 30 mL/min calculated by the Cockcroft-Gault formula or measured by 24-hour urine collection
13. Patients must meet the following cardiovascular parameters.

    1. Left ventricular ejection fraction (LVEF) ≥ 50 % by echocardiogram.
    2. QT interval with Fridericia correction method (QTcF) on screening electrocardiogram, defined as QTcF of ≤450 ms in males or ≤470 ms in females.
14. The effects of this agent on the developing human fetus are unknown. For this reason, and because other therapeutic agents used in this trial may be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 90 days after last treatment. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy #CLN1114; this applies to patients enrolled at MDA only. External participating sites will follow their own institutional policies/SOP.) This includes all female patients between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (follicle-stimulating hormone and estradiol in menopausal range, who have received whole pelvic radiation therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.
15. Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), tubal ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
16. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of treatment.
17. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patient has a white blood cell count > 10 x 10⁹/L. Hydroxyurea, and/or cytarabine (up to 2 g/m2 total) used as supportive care is permitted to meet this criterion.
2. Patients with known symptomatic or uncontrolled CNS leukemia.
3. Patient has systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate treatment.
4. Patients with the following cardiovascular conditions:

   1. Congestive heart failure, NYHA class ≥II, cardiomyopathy, active ischemia, or any other uncontrolled cardiac condition such as angina pectoris or myocardial infarction, clinically significant arrhythmia requiring therapy including anticoagulants within the past 6 months or at screening, (stable medical therapy for > 6 months is acceptable)
   2. Clinically significant uncontrolled hypertension at the time of screening,
   3. Patients with a history of documented pericarditis (any CTCAE grade) or pericardial effusions of at least CTCAE Grade 3 within 3 months before the start of treatment with MT-0169.
   4. Received chemotherapy with anthracycline agents at the doxorubicin equivalent cumulative dose (sum for all agents combined) of 450 mg/m2 body surface area, or a lower total doxorubicin equivalent cumulative dose that, in the opinion of the Investigator, would increase the risk of cardiomyopathy in this study.

   i. For patients who have received a cumulative dose of an anthracycline of more than 300 mg/m2 , approval must first be obtained from the Medical Monitor
5. Patients with a history of mediastinal irradiation.
6. Prior use of any cytotoxic chemotherapy, targeted therapy, antibody-drug conjugates, immunotherapy, or other investigational therapies within 2 weeks or 5 half-lives, whichever is shorter, prior to starting MT-0169. All prior therapy related toxicities should have resolved to grade ≤1.
7. Patients relapsing after allo-SCT may be eligible if they have recovered from all transplant-related toxicities and are off all immunosuppression, with no more than grade 1 chronic GVHD. Physiologic ("replacement") dose of steroids (≤10 mg prednisone or equivalent) may be acceptable. Patients must be off all immunosuppression, including calcineurin inhibitors, for at least 2 weeks or 5 half-lives, whichever is longer, prior to enrollment on study.
8. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection with detectable viral DNA or RNA, respectively, or known HIV infection.
9. Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator.
10. Any previous or concomitant malignancy, except when the patient has completed definitive curative-intent treatment with chemotherapy and/or surgery and/or radiotherapy at least 3 months prior to enrollment. Patients having completed definitive treatment for the following conditions may be eligible immediately after completion of definitive curative-intent therapy, after healing of wounds, and no evidence of residual disease by examination, imaging, and/or cytology/pathology, e.g., non-melanoma skin cancers, or a carcinoma in-situ, e.g., ductal carcinoma in situ, urothelial cancer, cervical cancer, localized prostate cancer, pre-cancerous colon polyp, etc.
11. Major surgery within 4 weeks prior to screening or a major wound that has not fully healed.
12. Patients under legal protection measure (guardianship, trusteeship or safeguard of justice) and/or uncontrolled psychiatric comorbidities, ongoing illicit substance abuse, inability, any impairment or unwillingness to comply with the treatments, follow-up, requirements and procedures of this clinical trial.
13. A known hypersensitivity or severe allergy to study drug components or diluents
14. Nursing women, women of childbearing potential (WOCBP) with positive urine or serum pregnancy test, or WOCBP who are not willing to maintain adequate contraception
15. Pregnant women are excluded from this study because study agents may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated on this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Maiti, MBBS, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org